CLINICAL TRIAL: NCT06583187
Title: Effect of Mandala Coloring on Fear, Anxiety, Emotional Symptoms and Postoperative Pain of Circumcised Children
Brief Title: Effect of Mandala Coloring of Circumcised Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Artvin Coruh University (Other)
Responsible Party: Principal Investigator, Gamze Akay, Assistant Professor, Artvin Coruh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Mandala Coloring
Record Dates: First submitted 2024-09-01; First posted 2024-09-03 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Circumcision
Keywords: anxiety; child; circumcision; emotional manifest; fear; pain; mandala painting
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Routine clinical care will be applied to the control group. No action will be taken.
- Experimental Group (Experimental): Before circumcision, the child will be coloring mandala pictures of the pediatric clinic.
  Interventions: Other: Coloring a mandala picture

INTERVENTIONS:
Other: Coloring a mandala picture — In the study, the experimental group was taken to their room on the day they came for circumcision and then had them paint mandalas. The coloring books chosen for mandala painting were determined to be appropriate for the age group of the children. The child was given a book and was given the freedom to paint the figures they wanted. Care was taken to ensure that the environment was quiet so that the child would be comfortable and calm. Care was taken to ensure that the crayons used in mandala painting did not contain carcinogenic substances and were anti-allergic.
  Arms: Experimental Group

SUMMARY:
The aim of this study was to determine the effect of mandala painting on fear, anxiety, emotional symptoms and postoperative pain of circumcised children.

DETAILED DESCRIPTION:
78 volunteer children between the ages of 6-12 who come for circumcision surgery will be randomly divided into two groups: mandala painting group and control group. Children will be evaluated before, during and after the procedure. Pain related to the circumcision procedure will be assessed using FLACC Pain Scale, fear will be assessed using High Fear Scale, anxiety will be assessed using Child Anxiety-State Scale and emotional state will be assessed using Emotional Indicators Scale. In addition, children's demographic data will be recorded in the Information Form.

ELIGIBILITY:
Inclusion Criteria:

Children between the ages of 6-12, Written and verbal consent given by their legal guardians, Can speak and are literate in Turkish, Have sufficient mental development to answer questions

Exclusion Criteria:

Children with congenital urological anomalies, Children with who did not agree to participate in the study and who were not in the specified age group

Ages: 6 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Male
Enrollment: 78 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Child Information Form | Baseline
  This form prepared by researchers in line with the literature, contains 13 questions regarding the child's age, previous hospitalization and surgery, information about the current surgery and who gave the information, the education level of the mother and father, the profession of the mother and father, the place of residence and economic status.

SECONDARY OUTCOMES:
The Wong-Baker Faces Pain Rating Scale | Baseline
  This scale was developed by Donna Wong and Connie Moran Baker in 1981. The scale is suitable for children between the ages of three and eighteen. The scale includes facial expressions that the child can enjoy and enjoy. For this reason, it has been stated that it gives more accurate results. The scale has scores of "0", "2", "4", "6", "8", and "10". "0" indicates no pain and "10" indicates the highest pain. This scale does not have a Cronbach alpha score. It has been reported that reliability studies have not been conducted on such scaling.

OTHER OUTCOMES:
Children's Fear Scale | Baseline
  The Children's Fear Scale (CFS) was used to assess procedural fear. The CFS is a reliable and valid tool for assessing procedural fear in school-aged children between the ages of 5 and 10 years.42 The CFS consists of five faces that are evenly distributed on a horizontal orientation. Each of them represents a different level of fear, the leftmost face marked as 0 and shows no fear, whereas the face on the far right marked as 4, shows the highest level of fear. The individuals reported their own fear levels by placing a mark on the horizontal axis. Before the procedure, the participating children were informed about the way of use of the scale. After the children stated that they understood how the scale can be used, they were asked to say how afraid they were. Children were asked a question as Can you look at these faces and choose the one which shows how afraid you are of having a circumcision? The mark was placed by each child was recorded.
Children's Emotional Manifestation Scale | Baseline
  The Children's Emotional Manifestation Scale (CEMS) was created in 2005 by Li & Lopez with the aim of offering a simple, objective and consistent method for nurses to determine the emotional behavior and anxiety of children during stressful medical procedures. The Turkish validity and reliability was performed by Çimke & Bayat in 2020. The scale measures emotional markers in children aged from 7 to 12 years undergoing operations. The scale examines 5 dimensions of facial expression, noises made by the child, activity, interaction and cooperation level of the child. Each item is rated from 1 to 5 points. As the points obtained on the scale increase, negative emotional manifestations increase. Assessment is from 5 to 25 points. The Turkish validity and reliability study for the scale found the Cronbach alpha value was 0.94.
Children's Anxiety State Scale | Baseline
  This scale was developed by Ersig et al. in 2013 measures the state anxiety of children aged 4-10 years. In 2017, Gerçeker et al. carried out Turkish validity study for the scale. CAS-S (State) is designed as a thermometer. At the bottom is the bulb chamber, and upwards are horizontal lines. Each horizontal line represents a score, and the thermometer has 10 points. The bulb chamber at the bottom is 0 points and indicates that there is no anxiety. It is interpreted as the rise of anxiety as it rises upwards. The peak is worth 10 points and refers to the highest anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice OĞUZHAN, Lecturer, Study Chair — Gümüşhane Universıty
Locations (1):
- Gümüşhane Hospital Pediatric Clinic, Gümüşhane, Turkey (Türkiye)

REFERENCES:
- [Background] Yeniay D, Tamdo An L, Yucak Ozdemir A, Ak An LO, Kay R SU. Effects of Videos and Therapeutic Music on Preoperative Anxiety and Postoperative Anxiety and Pain Levels in Boys Who Undergo Circumcision. J Perianesth Nurs. 2023 Dec;38(6):918-924. doi: 10.1016/j.jopan.2023.04.007. Epub 2023 Aug 16. PMID 37589631